CLINICAL TRIAL: NCT03106610
Title: A Pilot Trial of Anti-PD-1 (Nivolumab) in Bladder Cancer Patients Recently Treated With Intravesical BCG Immunotherapy
Brief Title: Trial of Anti-PD-1 (Nivolumab) in Bladder Cancer Patients Recently Treated With Intravesical BCG Immunotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0432; NCI-2017-00647 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-03-30; First posted 2017-04-10 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Cancer of urothelium; Transitional cell carcinoma; Carcinoma in situ; Nivolumab; BMS-936558; Opdivo; Questionnaires; Surveys
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Carcinoma in Situ | interventions — Nivolumab; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Participants receive Nivolumab by vein over about 60 minutes on Day 1 of Cycles 1-3 before scheduled surgery. Each study cycle is 14 days (2 weeks).
  Questionnaires completed on Day 1 of Cycles 1-3, at the visit before surgery, and 4 weeks after surgery.
  Interventions: Drug: Nivolumab; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Nivolumab — 3 mg/kg of body weight by vein over about 60 minutes on Day 1 of Cycles 1-3.
  Other Names: BMS-936558; Opdivo
Behavioral: Questionnaires — 2 quality-of-life questionnaires completed on Day 1 of Cycles 1-3, at the visit before surgery, and 4 weeks after surgery.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to learn about the tolerability of nivolumab in patients who have bladder cancer, were previously treated with BCG immunotherapy, and who have a cystectomy (removal of all or part of the bladder) scheduled as part of their standard care.

This is an investigational study. Nivolumab is FDA approved and commercially available to treat metastatic (has spread) melanoma or non-small cell lung cancer (NSCLC) after the disease has gotten worse while receiving platinum-based chemotherapy. The use of nivolumab in this study is considered investigational.

Up to 10 participants will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

Each study cycle is 14 days (2 weeks).

If you are found to be eligible to take part in this study, you will receive nivolumab by vein over about 60 minutes on Day 1 of Cycles 1-3.

Length of Study:

You may receive nivolumab for up to 3 cycles before your scheduled surgery. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits (described below).

Study Visits

On Day 1 of Cycles 1-3 and at the visit before your surgery:

* You will have a physical exam.
* Blood (about 3-4 teaspoons) will be drawn for routine tests.
* You will be asked to complete 2 quality-of-life questionnaires. These will take about 10 minutes to complete.
* If you can become pregnant, urine or part of the above routine blood sample will be used for a pregnancy test.

Surgery (Cystectomy):

About 8 weeks after you join the study, you will have surgery for bladder cancer. You will sign a separate consent form that describes the surgery and its risks.

Follow Up:

About 4 weeks after surgery:

* You will have a physical exam.
* Blood (about 3-4 teaspoons) will be drawn for routine tests.
* You will be asked to complete the 2 quality-of-life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Patients included in the study must be >/= 18 years old.
2. Histological or cytological evidence of transitional cell carcinoma or carcinoma in situ of the urothelium involving the bladder or prostatic urethra following treatment with BCG with the recommendation to proceed for cystectomy. Minor histologic variants (< 50% overall) are acceptable. Diagnosis must be within 1 year of study entry.
3. Patent must have BCG unresponsive non-muscle-invasive bladder cancer defined as: Persistent or recurrence of CIS within 12 months, or recurrence of CIS with Ta/T1 papillary disease within 12 months, or recurrence of high grade Ta or T1 papillary disease alone within 6 months of receiving at least two courses of intravesical BCG (at least five of six induction doses and at least two doses of either a maintenance course of BCG or a 2nd re-induction of BCG; or T1 high-grade disease at the first evaluation following induction of BCG alone (at least five of six induction doses).
4. Subjects must have received intravesical treatment with at least two doses of BCG within six months of nivolumab treatment initiation.
5. Evaluable tumor tissue (archived or new biopsy) must be available for pre-treatment biomarker analysis and baseline immune monitoring studies
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
7. Screening laboratory values must meet the following criteria and must be obtained within 14 days prior to first dose: a) WBC >/= 2000/µL; b) Neutrophils >/= 1500/µL; c) Platelets >/= 100 x 10^3/mcl; d) Hemoglobin >/= 9.0 g/dL; e) AST and ALT </= 3 x ULN; f) Total Bilirubin </= 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
8. Inclusion 6) continued; g.Serum creatinine </=1.5 x ULN or creatinine clearance (CrCl) >/=30 mL/min (using the Cockcroft-Gault formula): 1) Female CrCl = (140 - age in years) x weight in kg x 0.85 / 72 x serum creatinine in mg/dL; 2) Male CrCl = (140 - age in years) x weight in kg x 1.00 / 72 x serum creatinine in mg/dL
9. Ability to understand and willingness to sign a written informed consent document.
10. Females of childbearing potential who are sexually active with a non-sterilized male partner and non-sterilized males must use a highly effective method of contraception for 28 days prior to the first dose of investigational product, and must agree to continue using such precautions for 180 days after the final dose of investigational product; cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. They must also refrain from egg cell donation for 180 days after the final dose of investigational product;
11. Inclusion 9) continued; a) Females of childbearing potential are defined as those who are not surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause)
12. Inclusion 9) continued; b) A highly effective method of contraception is defined as one that results in a low failure rate (ie, less than 1% per year) when used consistently and correctly. The acceptable methods of contraception are: Barrier Method (e.g. male condom with spermicide, copper T intrauterine device, or levonorgestrel-releasing intrauterine system - Mirena®) or Hormonal Methods (e.g. implants, hormone shot or injection, combined pill, minipill, or patch).

Exclusion Criteria:

1. Patients with high risk muscle invasive urothelial carcinoma (hydronephrosis, palpable mass on examination under anesthesia,muscle invasive urothelial carcinoma with lymphovascular invasion on pathologic specimen, >T3 disease) or those with lymph node positive or metastatic disease are to be excluded.
2. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
3. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, prostate cancer without evidence of PSA progression or carcinoma in situ such as the following: gastric, prostate, cervix, colon, melanoma, or breast for example.
4. Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
5. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
6. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4) antibody, anti-CD137, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
7. All toxicities attributed to prior anti-cancer therapy other than neuropathy, alopecia and fatigue must have resolved to Grade 1 (NCI CTCAE version 4) or baseline before administration of study drug. Subjects with toxicities attributed to prior anti-cancer therapy which are not expected to resolve and result in long lasting sequelae, such as neuropathy after platinum based therapy, are permitted to enroll. Neuropathy must have resolved to Grade 2 (NCI CTCAE version 4).
8. Treatment with any chemotherapy, radiation therapy, biologics for cancer, or investigational therapy within 28 days of first administration of study treatment.
9. Physical and Laboratory Test Findings; a) Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (RNA) or hepatitis C antibody (HCV antibody) indicating acute or chronic infection; b) Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
10. Allergies and Adverse Drug Reaction; a) History of allergy to study drug components; b) History of severe hypersensitivity reaction to any monoclonal antibody.
11. Sex and Reproductive Status; a) Women of childbearing potential (WOCBP) who are pregnant or breastfeeding; b) Women with a positive pregnancy test at enrollment or prior to administration of study medication
12. Prisoners or subjects who are involuntarily incarcerated
13. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Safety of Nivolumab in Subjects Previously Treated with Intravesical Bacillus Calmette-Guerin (BCG) Immunotherapy assessed per NCI CTCAE version 4 | 12 weeks
  Safety assessed per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.

SECONDARY OUTCOMES:
Tolerability of Nivolumab in Subjects Previously Treated with Intravesical Bacillus Calmette-Guerin (BCG) Immunotherapy assessed using AUASS | 12 weeks
  Tolerability assessed by measurement of local urinary symptoms using the American Urological Association Symptom Score (AUASS).
Systemic Symptom Burden of Nivolumab in Subjects Previously Treated with Intravesical Bacillus Calmette-Guerin (BCG) Immunotherapy assessed using MDASI | 12 weeks
  Systemic symptom burden assessed using the MD Anderson Symptom Inventory (MDASI).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Campbell, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org